CLINICAL TRIAL: NCT04228133
Title: Home-Delivered Attention Control Training for Post Traumatic Stress Disorder: A Randomized Controlled Trial
Brief Title: Home-Delivered Attention Control Treatment for Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor of Psychology and Neuroscience School of Psychological Sciences Sagol School of Neuroscience Tel Aviv University, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAU-ACT
Record Dates: First submitted 2020-01-01; First posted 2020-01-14 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: PTSD
Keywords: PTSD; attention training; cognitive bias modification; home-delivered intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-delivered attention control training (ACT) (Experimental): A home-delivered ACT comprised of 8 sessions with a variation of the dot-probe task in which the target probe replaces the neutral and threat stimuli with an equal probability to reduce attention bias variability (ABV).
  Interventions: Behavioral: Attention Control Training (ACT)
- Home-delivered attention bias modification (ABM) (Placebo Comparator): A home-delivered ABM comprised of 8 sessions with a variation of the dot-probe task in which the target probe always replaces the threat stimuli to induce diversion of attention away from threat.
  Interventions: Behavioral: Attention Bias Modification (ABM)

INTERVENTIONS:
Behavioral: Attention Control Training (ACT) — A home-delivered version of ACT will be administered in this study. ACT will be comprised of 8 sessions with a variation of the dot-probe task in which the target probe replaces the neutral and threat stimuli with an equal probability to reduce attention bias variability (ABV). In addition, sessions will include video conference with the experimenter. This condition has found to be more effective in PTSD symptom reduction compared to ABM.
  Arms: Home-delivered attention control training (ACT)
Behavioral: Attention Bias Modification (ABM) — A home-delivered version of ABM will be administered in this study. ABM will be comprised of 8 sessions with a variation of the dot-probe task in which the target probe always replaces the threat stimuli to induce diversion of attention away from threat. In addition, sessions will include video conference with the experimenter. This condition has found to be have an inferior effect on PTSD symptom reduction compared to ACT, and thus, this ABM condition has been chosen as a control condition.
  Arms: Home-delivered attention bias modification (ABM)

SUMMARY:
The aim of the study is to explore the efficacy of home-delivered Attention Control Training (ACT) for Posttraumatic Stress Disorder (PTSD).

Three randomized controlled trials have shown that attention bias modification protocols applying attention control training (ACT) aimed to balance attention between threat-related and neutral stimuli are efficient in reducing PTSD symptoms. However, contrary to in-clinic administration, such as applied in the above mentioned studies, home-delivered attention bias modification was not effective in reducing symptoms among treatment-seeking patients.

It is crucial to continue examining the efficacy of home-delivered ACT as PTSD entails functional impairments that might impede treatment-seeking patients from reaching to clinics to receive treatment. This could also inform other ABM protocols designated to treat other disorders.

DETAILED DESCRIPTION:
The aim of the study is to explore the efficacy of home-delivered Attention Control Training (ACT) for Posttraumatic Stress Disorder (PTSD).

Three randomized controlled trials have shown that attention bias modification (ABM) protocols applying attention control training (ACT) aimed to balance attention between threat-related and neutral stimuli are efficient in reducing PTSD symptoms. However, contrary to in-clinic administration, such as applied in the above mentioned studies, home-delivered ABM was not effective in reducing symptoms among treatment-seeking patients.

It is crucial to continue examining the efficacy of home-delivered ACT as PTSD entails functional impairments that might impede treatment-seeking patients from reaching to clinics to receive treatment. This could also inform other ABM protocols designated to treat other disorders.

To overcome some critical differences between home and lab environments, the investigators developed a home-delivered ACT protocol that resembles as much as possible the typical-in-lab protocol. Specifically, participants will be accompanied during their training sessions using internet-based video conference, permitting a better control for the physical environment before and during the session and a direct interaction with the experimenters.

To test its efficacy, the investigators will recruit participants that are diagnosed with PTSD and will be randomly assigned to one of two home-delivered conditions: ACT and a control ABM condition. It is hypothesized that home-delivered ACT will produce greater reduction in PTSD symptoms relative to a control ABM protocol. It is also expected that ACT will reduce attention bias variability to a greater extent compared to the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Meeting a current diagnosis of Post-Traumatic Stress Disorder (PTSD) according to DSM-V (American Psychiatric Association, 2013);
* Having a home PC with internet access, web cam, microphone and speakers. Operation system must be windows 7 or a newer version.

Exclusion Criteria:

* A diagnosis of psychotic or bipolar disorders.
* A diagnosis of a neurological disorder (i.e., epilepsy, brain injury).
* Suicidal ideation.
* Drugs or alcohol abuse.
* Non-fluent Hebrew.
* A pharmacological or psychotherapy treatment that is not stabilized in the past 3 months (a stable treatment will not be a reason for exclusion from the study).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the total severity score of the CAPS-5 interview | up to 2 weeks pre-treatment and 1-2 weeks post-treatment
  The Clinician Administered PTSD Scale (CAPS-5), is a structured interview that will be used to make a diagnosis of PTSD according to the DSM-V criteria. This interview is consists of 30 items regarding the frequency and intensity of PTSD symptoms and a total score of severity is been rated, with higher scores denoting higher symptom severity.

SECONDARY OUTCOMES:
Change from baseline of the total score of the PTSD Checklist (PCL-5) | up to 2 weeks pre-treatment and 1-2 weeks post-treatment
  The PCL-5, is a 20-item National Center for PTSD Checklist of the Department of Veterans Affairs. Scores can range from 0 to 80, with higher scores reflecting more symptoms of PTSD.

OTHER OUTCOMES:
Change from baseline of the total score of the PHQ-9 | up to 2 weeks pre-treatment and 1-2 weeks post-treatment
  The PHQ-9 is a 9-item scale for depression symptoms (Kroenke, Spitzer, & Williams, 2001). Scores can range from 0 to 27, with higher scores reflecting more symptoms of depression.
The Credibility/Expectancy Questionnaire (CEQ) | up to 2 weeks pre-treatment and 1-2 weeks post-treatment
  The Credibility/Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000). This instrument consists of 6 items which derive two factors: expectancy for change and treatment credibility. This CEQ will be used to explore whether expectancies or treatment credibility are related to outcomes. It demonstrated high internal consistency and good test-retest reliability.
The CGI/S | up to 2 weeks pre-treatment and 1-2 weeks post-treatment
  Severity and improvement scales (CGI-S/I) will be used to assess participants global clinical condition. The CGI-S and the CGI-I are single-items, clinician-reported, measure assessing severity and improvement of illness using a 7-point Likert-type scale. The CGI-S/I has good inter-rater reliability and concurrent validity with other measures. This tool is widely used in clinical trials concerning psychopathology treatments and has good sensitivity to clinical change.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badura-Brack AS, Naim R, Ryan TJ, Levy O, Abend R, Khanna MM, McDermott TJ, Pine DS, Bar-Haim Y. Effect of Attention Training on Attention Bias Variability and PTSD Symptoms: Randomized Controlled Trials in Israeli and U.S. Combat Veterans. Am J Psychiatry. 2015 Dec;172(12):1233-41. doi: 10.1176/appi.ajp.2015.14121578. Epub 2015 Jul 24. PMID 26206075
- [Background] Lazarov A, Suarez-Jimenez B, Abend R, Naim R, Shvil E, Helpman L, Zhu X, Papini S, Duroski A, Rom R, Schneier FR, Pine DS, Bar-Haim Y, Neria Y. Bias-contingent attention bias modification and attention control training in treatment of PTSD: a randomized control trial. Psychol Med. 2019 Oct;49(14):2432-2440. doi: 10.1017/S0033291718003367. Epub 2018 Nov 12. PMID 30415648
- [Background] Linetzky M, Pergamin-Hight L, Pine DS, Bar-Haim Y. Quantitative evaluation of the clinical efficacy of attention bias modification treatment for anxiety disorders. Depress Anxiety. 2015 Jun;32(6):383-91. doi: 10.1002/da.22344. Epub 2015 Feb 24. PMID 25708991
- [Background] Hedges DW, Brown BL, Shwalb DA. A direct comparison of effect sizes from the clinical global impression-improvement scale to effect sizes from other rating scales in controlled trials of adult social anxiety disorder. Hum Psychopharmacol. 2009 Jan;24(1):35-40. doi: 10.1002/hup.989. PMID 18980264
- [Background] Kadouri A, Corruble E, Falissard B. The improved Clinical Global Impression Scale (iCGI): development and validation in depression. BMC Psychiatry. 2007 Feb 6;7:7. doi: 10.1186/1471-244X-7-7. PMID 17284321
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729